CLINICAL TRIAL: NCT02441920
Title: Chronic Periodontitis and Tooth Loss in Patients With Rheumatoid Arthritis
Status: Terminated | Type: Observational
Why Stopped: Incomplete student research project
Sponsor: University of Birmingham (Other)
Collaborators: Dudley Group NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RG_09-196
Record Dates: First submitted 2015-05-08; First posted 2015-05-12 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2017-02

CONDITIONS: Periodontitis; Rheumatoid Arthritis
MeSH Terms: conditions — Periodontitis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with rheumatoid arthritis: The inception cohort of 400 patients will be followed up for 20 years following recruitment.

SUMMARY:
Periodontitis is a highly prevalent chronic inflammatory disease that is characterized by loss of the periodontal ligament and alveolar bone, and is a major cause of tooth loss. Results from clinical and epidemiological studies have suggested that periodontitis and tooth loss are more prevalent in individuals with rheumatoid arthritis (RA). There is evidence to suggest that periodontitis could indeed be a causal factor in the initiation and maintenance of the autoimmune inflammatory response that occurs in RA. If so, chronic periodontitis might represent an important modifiable risk factor for RA. However, to date longitudinal studies on the effect of periodontitis on disease progression in RA are lacking. The aim of the present study is to assess the periodontal status of patients enrolled in an established longitudinal cohort of RA patients. These data will then be analysed to evaluate whether or not periodontal inflammation is related to parameters of rheumatoid arthritis.

DETAILED DESCRIPTION:
Chronic periodontitis is arguably the most prevalent chronic inflammatory disease in humans. The defining feature of periodontitis is chronic inflammation of the tooth-supporting tissues, leading to the progressive destruction of periodontal ligament and alveolar bone. Periodontitis is a very common disease, affecting over 30% of adults aged 65 years or above in the UK. Results from a growing number of clinical studies point towards a potential association between chronic periodontitis and systemic rheumatic diseases- in particular, rheumatoid arthritis (RA). If proven, such an association would be very important from a clinical and public health perspective for several reasons. First, there are several processes through which chronic periodontitis might be part of a causal pathway in the pathogenesis and/or disease activity status of RA. Given the high prevalence of chronic periodontitis, a large proportion of the incidence and/or morbidity of RA could be attributable to chronic periodontitis, if causality was confirmed.

Importantly, chronic periodontitis would represent a modifiable risk factor, as effective treatments for this disease are available. Second, chronic periodontitis would contribute to morbidity in patients with RA even if the association was noncausal. Periodontitis is a leading cause of tooth loss in adults, which can have important clinical consequences, including impaired nutritional status and quality of life. Furthermore, chronic periodontitis is associated with an increased incidence of coronary heart disease and stroke, and emerging evidence indicates that this association might, in part, be causal, and thus periodontitis may contribute to the increased cardiovascular morbidity and mortality in RA.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilling the 1987 revised criteria for the classification of Rheumatoid arthritis
* Under active follow-up by a rheumatologist at the Dudley Group of Hospitals
* Participation in study 04/Q2702/18 "Establishment of an inception cohort for the prospective evaluation of predictors of cardiovascular morbidity and mortality in patients with rheumatoid arthritis".
* Participation in study 04/Q2702/18 "A prospective study of micro and macro vascular disease in a cohort of patients with Rheumatoid arthritis").
* Written informed consent

Exclusion Criteria:

* No absolute exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have already consented to their participation in a co-existing study will be eligible for inclusion: 04/Q2702/18 submitted 08/06/ 2004 "Establishment of an inception cohort for the prospective evaluation of predictors of cardiovascular morbidity and mortality in patients with rheumatoid arthritis."
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2010-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Associations between periodontal parameters and RA related factors including disease activity, severity, progression, and comorbidities | 1 year
  incomplete student research project

CONTACTS AND LOCATIONS:
Overall Officials: Paola de Pablo, Principal Investigator — University of Birmingham